# INFORMED CONSENT WITH HIPAA AUTHORIZATION TO COLLECT, USE, AND DISCLOSE PROTECTED HEALTH INFORMATION (PHI)

## A PHASE I/II CLINICAL TRIAL OF PEPCAN IN HEAD AND NECK CANCER PATIENTS IN REMISSION TO REDUCE RECURRENCE REGARDLESS OF HPV STATUS

| Subject Name: | |
|---|---|
| Subject MRN: | |
| Principal Investigator: | Omar Atiq, MD Professor of Medicine and Otolaryngology - Head and Neck Surgery Winthrop P. Rockefeller Cancer Institute, College of Medicine, University of Arkansas for Medical Sciences 4301 W. Markham St., Slot 508 Little Rock, AR 72205 (501) 686-8530 or after hours at (501) 686-6080 |
| Sub-Investigators: | Mayumi Nakagawa, MD, PhD<br>Professor, Dept. of Pathology, College of Medicine<br>University of Arkansas for Medical Sciences |
| | Konstantinos Arnaoutakis, MD, FACP<br>Associate Professor of Medicine, Hematology-Oncology<br>College of Medicine<br>University of Arkansas for Medical Sciences |
| | Mauricio Moreno, MD<br>Associate Professor, Dept. of Otolaryngology - Head & Neck Surgery<br>University of Arkansas for Medical Sciences |
| | Emre Vural, MD, FACS Professor and Attending Surgeon, Dept. of Otolaryngology - Head & Neck Surgery University of Arkansas for Medical Sciences |
| | Jumin Sunde, MD<br>Assistant Professor, Dept. of Otolaryngology - Head & Neck Surgery<br>University of Arkansas for Medical Sciences |
| | Gary Lewis, MD Assistant Professor, Dept. of Radiation Oncology University of Arkansas for Medical Sciences |


University of Arkansas for Medical Sciences

Samantha Rose, APRN ICE CASL CA Clinical Staff

Medical Monitor: Rangaswamy Govindarajan, MD

Professor, Dept. Internal Medicine, Hematology-Oncology

College of Medicine

University of Arkansas for Medical Sciences

Study Statistician: Horace (Trey) Spencer

Biostatistics Project Manager, Dept. Biostatistics

College of Medicine

University of Arkansas for Medical Sciences

Sponsor: University of Arkansas for Medical Sciences (UAMS)

Funding Source: UAMS/National Institutes of Health (National Cancer Institute)

Study Location: UAMS Winthrop P. Rockefeller Cancer Institute (WPRCI)

Phone Numbers: (501) 686-8530 or after hours at (501) 686-6080, Dr. Atiq

## KEY INFORMATION FOR A PHASE I/II CLINICAL TRIAL OF PEPCAN IN HEAD AND NECK CANCER PATIENTS IN REMISSION TO REDUCE RECURRENCE REGARDLESS OF HPV STATUS:

We are asking you to choose whether or not to volunteer for a research study using an investigational new vaccine, called PepCan, to try to reduce the recurrence of head and neck cancer in subjects who are in complete remission (free from the evidence of cancer).

This section is to give you key information to help you decide whether or not to participate. We have included detailed information after this section. Ask the research team questions. If you have questions later, the contact information for the research investigator in charge of the study is below.

#### WHAT IS THE STUDY ABOUT AND HOW LONG WILL IT LAST?

This study examines use of a vaccine called PepCan for subjects who have completed treatment for head and neck cancer. By doing this study, we hope to learn whether the vaccine is safe. In addition, we will look at how well the vaccine works in reducing cancer recurrence [cancer coming back again] and how your body's immune system responds to the vaccine. Your participation in this research will last about two years. Some subjects will receive the vaccine, and some will receive a placebo (salt water, with no medicine in it). If you join the study, you will be asked to:

- attend 10 required study visits
- optional follow-up visits as needed,
- provide four (4) saliva samples and stool samples for the research,
- provide four (4) blood samples for the research,
- receive a total of seven (7) injections of the PepCan vaccine or placebo (salt water). You will have a 3 out of 4 chance of receiving the PepCan vaccine.

The purpose of this research is to gather information on the safety and effectiveness of a new therapeutic HPV vaccine, called PepCan. This new vaccine is not approved by the United States Food and Drug Administration (FDA). The vaccine consists of a laboratory-made piece of HPV protein called E6 and yeast extract called Candin®.

#### WHY MIGHT I CHOOSE TO VOLUNTEER FOR THIS STUDY?

You have been invited to be screened for this study because you have been diagnosed with head and neck cancer and have achieved complete remission. Your participation in the study will contribute toward the development of this new vaccine and it is possible that it may reduce your chances of your cancer returning. For a complete description of benefits refer to the Full Consent.

## WHY MIGHT I CHOOSE NOT TO VOLUNTEER FOR THIS STUDY?

You may not wish to participate in the study as there may be no direct benefit for you. This means the vaccine may not prevent your cancer from returning or you may be in the group that does not receive the vaccine. There may be some side effects such as injection-site reactions (redness, itching, swelling), nausea, flu-like syndrome, fever, headache, chills, and muscle aches. There will be no compensation provided for your participation. Research information collected during the study is not considered standard of care and, therefore, will not be released to you. For a complete description of benefits refer to the Full Consent.

Standard-of-care alternative treatments may also be available. For a complete description of alternate treatment/procedures ask your doctor.

Sponsor: UAMS

#### WILL IT COST ME ANYTHING TO BE IN THIS STUDY?

You and/or your health insurance will be required to pay for those services, supplies, procedures and care that you continue to require for your routine medical care during this study (meaning the procedures and services you would have had even if you were not in the study). You will be responsible for any co-payments and/or deductibles as required by your insurance for such routine medical care. Occasionally, insurance may not cover standard of care procedures for people are enrolled in a research study. If you have any questions about costs to you that may result from taking part in the research, please speak with the study doctors and study staff. If necessary, we will arrange for you to speak with someone in the University of Arkansas for Medical Sciences Patient Financial Services about these costs.

#### DO I HAVE TO TAKE PART IN THE STUDY?

No. It is okay to say no. If you decide to take part in the study, it should be because you really want to volunteer. You will not lose any services, benefits, or rights you would normally have if you choose not to volunteer.

If you are a student or employee, nothing about your education or employment will change no matter what you decide.

## WHAT IF I HAVE QUESTIONS, SUGGESTIONS, OR CONCERNS?

You can contact the person in charge of the study. Dr. Omar Atig in the UAMS College of Medicine, with any questions, suggestions, or concerns at (501) 686-8530 or after hours at (501) 686-6080.

If you have any questions, suggestions, or concerns about your rights as a volunteer in this study, or wish to speak to someone not directly involved in the research, you can call the UAMS Institutional Review Board (IRB) at 501-686-5667 during business hours.

If you want to know more about the research, let the study team know so they can give you more information.

Also, tell the study team if you have decided you don't want to be in the study. It is perfectly okay to say no.


#### INTRODUCTION

This is clinical trial, a type of research study, being conducted at the University of Arkansas for Medical Sciences (UAMS). Participants in the study will be men and women aged 18 years or older who have recently had head and neck cancer. Up to 150 men and women will be enrolled into the study for screening, and 100 eligible men and women will receive 7 injections of the vaccine PepCan or placebo (salt water). You will be assigned by chance, like flipping a coin to receive either PepCan or placebo. Your chances of receiving PepCan will be 3 times as much as receiving placebo. You and the study staff (except for the pharmacists) will not know which injection you receive until after the study has been completed. The first 4 doses of the PepCan vaccine or placebo (salt water) will be given once every 3 weeks. Then, the remaining 3 doses of the PepCan vaccine or placebo (salt water) will be given once every 3 months. HPV stands for human papillomavirus, and it can cause certain cancers (including head and neck cancer) and warts. Participants in this research study are not at risk of getting HPV as a result of receiving the vaccine since it contains synthetically (artificially) made fragments of HPV.

#### WHO CAN PARTICIPATE IN THIS STUDY?

In order to qualify to take part in the study, you must be at least 18 years of age, have received treatments (surgery, radiation, and/or chemotherapy) for head and neck cancer in the last 120 days, currently have no evidence of disease, be able to perform routine everyday tasks at home independently, and have blood pressure, heart rate, breathing rate, and temperature within certain ranges (a study staff member will review these in detail with you at the Screening Visit).

You will not be able to participate in the study, if you are pregnant or plan to become pregnant, are breastfeeding, are allergic to yeast, have been to the emergency room/have been hospitalized for asthma, have received PepCan in the past, have had recurrence of head and neck cancer, and/or if investigators believe that it is not in your best interest to participate in the study. Your white blood cell and red blood cell counts would also need to be in certain ranges when tested at the Screening Visit (a study staff member will review these with you in detail).

#### **WHAT WILL HAPPEN**

- We will ask you a series of questions to see if you qualify for the study.
- After the study has been explained to you and if you agree to participate, you will be asked to provide informed consent.
- You'll be asked to provide your name, date of birth, ethnicity, and contact information, so that UAMS may make an appointment for you.
- A Screening Visit appointment will be made in the UAMS Winthrop P. Rockefeller Cancer Institute (WPRCI)

## **Screening Visit (UAMS Winthrop P. Rockefeller Cancer Institute)**

- You'll be asked to fill out the "Subject Contact Information" form, which will gather
  information such as your name, date of birth, phone numbers, e-mail address, mailing
  address, race, and ethnicity.
- You'll be asked to provide medical history including drug allergies and current medications.
- You'll be asked to complete the Screening Visit Questionnaire. You will be asked to fill out
  a form regarding your use of nicotine and alcohol, your employment, your sexual history,
  and your motivations for joining the study.
- Vital signs will be obtained and a physical examination will be performed.

Sponsor: UAMS

- Women of childbearing potential will be asked to take a urine pregnancy test.
- The risks involved with becoming pregnant will be discussed with women of childbearing potential and they will be asked to specify which birth-control method they will use during the study.
  - Examples of ways you can prevent getting pregnant include pills, patches, rings, implants, shots, double-barrier methods (condoms and spermicide), abstinence, or vasectomies of your male partner combined with another birth-control method.
- About 1 tablespoon of blood will be drawn for clinical testing. Results from standard of care blood tests may be used within 30 days prior to the date the consent form is signed.
- You will be asked to swish a tablespoon of mouthwash for at least 30 seconds in your mouth and spit it into a specimen cup. You should not have brushed for 2 hours and eaten for 10 minutes before doing so.
- You will be asked to complete a questionnaire about antibiotic usage.
  - You will be asked to provide a stool sample after you return home and will be given another questionnaire asking about antibiotic usage, packaging instructions and shipping supplies to send the sample back to UAMS.

If all results and information are not available during the screening visit, you will be contacted later by study staff as to whether you are eligible for vaccination. If you are eligible, Vaccination Visits will be scheduled after you returned the stool sample. Visit 1 will be scheduled within 90 days of the screening visit. If you are not eligible, you will not need to provide a stool sample and you may discard the kit. A physician or nurse will provide instructions about standard follow-up care.

## Visit 1 (after receiving stool sample back; UAMS Winthrop P. Rockefeller Cancer Institute)

- You'll be asked about any medication changes.
- Women of childbearing potential will be asked to take a urine pregnancy test.
- Eight to ten tubes of blood (up to 7 tablespoons total) will be drawn for clinical and immunology testing. Additional tubes may be drawn for standard of care.
  - The blood may be used to study how your white cells are reacting to HPV, to allow them to grow in a laboratory, for tissue (HLA) typing, genetic testing of your immune cells and related genes, and other similar tests. In addition, the blood may be used for other testing to see if the vaccine worked in your body by examining proteins and other types of specialized cells.
- Vital signs will be obtained before vaccine injection.
- PepCan vaccine or placebo (salt water) will be injected under your skin in either one of your arms or one of your legs.
- After resting for at least 30 min after the injection, vital signs will be obtained.
- You'll be offered a dose of ibuprofen or naproxen (e.g., Advil® or Aleve®). You do not have to take it, but it might help limit possible reactions that may occur.

## Visit 2 (3 weeks after Visit 1; UAMS Winthrop P. Rockefeller Cancer Institute)

- You'll be asked if you experienced any side effects or reactions to the last vaccination.
- You'll be asked about any medication changes.
- Women of childbearing potential will be asked to take a urine pregnancy test.
- Vital signs will be obtained before vaccine injection.


- PepCan vaccine or placebo (salt water) will be injected under your skin in either one of your arms or one of your legs.
- After resting for at least 30 min after the injection, vital signs will be obtained.
- You'll be offered a dose of ibuprofen or naproxen. You do not have to take it, but it might help limit possible reactions that may occur.

## Visit 3 (3 weeks after Visit 2; UAMS Winthrop P. Rockefeller Cancer Institute)

- You'll be asked if you experienced any side effects or reactions to the last vaccination.
- You'll be asked about any medication changes.
- Women of childbearing potential will be asked to take a urine pregnancy test.
- About 1 tablespoon of blood will be drawn for clinical testing.
- Vital signs will be obtained before vaccine injection.
- PepCan vaccine or placebo (salt water) will be injected under your skin in either one of your arms or one of your legs.
- After resting for at least 30 min after the injection, vital signs will be obtained.
- You'll be offered a dose of ibuprofen or naproxen. You do not have to take it, but it might help limit possible reactions that may occur.

## Visit 4 (3 weeks after Visit 3; UAMS Winthrop P. Rockefeller Cancer Institute)

- You'll be asked if you experienced any side effects or reactions to the last vaccination.
- You'll be asked about any medication changes.
- Women of childbearing potential will be asked to take a urine pregnancy test.
- Vital signs will be obtained before vaccine injection.
- PepCan vaccine or placebo (salt water) will be injected under your skin in either one of your arms or one of your legs.
- After resting for at least 30 min after the injection, vital signs will be obtained.
- You'll be offered a dose of ibuprofen or naproxen. You do not have to take it, but it might help limit possible reactions that may occur.

## Visit 5 (3 months after Visit 4; UAMS Winthrop P. Rockefeller Cancer Institute)

- You'll be asked if you experienced any side effects or reactions to the last vaccination.
- You'll be asked about any medication changes.
- Women of childbearing potential will be asked to take a urine pregnancy test.
- You will be asked to swish approximately one tablespoon of mouthwash for at least 30 seconds in your mouth and spit it into a specimen cup. You should not have brushed for 2 hours and eaten for 10 minutes before doing so.
  - o You will be asked to complete a questionnaire about antibiotic usage.
- Eight to ten tubes of blood (up to 7 tablespoons total) will be drawn for clinical and immunology testing. Additional tubes may be drawn for standard of care.
  - The blood may be used to study how your white cells are reacting to HPV, to allow them to grow in a laboratory, for tissue (HLA) typing, genetic testing of your immune cells and related genes, and other similar tests. In addition, the blood may be used for other testing to see if the vaccine worked in your body by examining proteins and other types of specialized cells.
- A physical exam will be performed.


Sponsor: UAMS

- Vital signs will be obtained before vaccine injection.
- PepCan vaccine or placebo (salt water) will be injected under your skin in either one of your arms or one of your legs.
- After resting for at least 30 min after the injection, vital signs will be obtained.
- You'll be offered a dose of ibuprofen or naproxen. You do not have to take it, but it might help limit possible reactions that may occur.
- You will be given a stool collection kit with another questionnaire asking about antibiotic usage, instructions and shipping supplies to send the sample back to UAMS.

## Visit 6 (3 months after Visit 5; UAMS Winthrop P. Rockefeller Cancer Institute)

- You'll be asked if you experienced any side effects or reactions to the last vaccination.
- You'll be asked about any medication changes.
- Women of childbearing potential will be asked to take a urine pregnancy test.
- About 1 tablespoon of blood will be drawn for clinical testing.
- A physical exam will be performed.
- Vital signs will be obtained before vaccine injection.
- PepCan vaccine or placebo (salt water) will be injected under your skin in either one of your arms or one of your legs.
- After resting for at least 30 min after the injection, vital signs will be obtained.
- You'll be offered a dose of ibuprofen or naproxen. You do not have to take it, but it might help limit possible reactions that may occur.

## Visit 7 (3 months after Visit 6; UAMS Winthrop P. Rockefeller Cancer Institute)

- You'll be asked if you experienced any side effects or reactions to the last vaccination.
- You'll be asked about any medication changes.
- Women of childbearing potential will be asked to take a urine pregnancy test.
- You will be asked to swish a tablespoon of mouthwash for at least 30 seconds in your mouth and spit it into a specimen cup. You should not have brushed for 2 hours and eaten for 10 minutes before doing so.
  - You will be asked to complete a questionnaire about antibiotic usage.
- About 1 tablespoon of blood will be drawn for clinical testing.
- A physical exam will be performed.
- Vital signs will be obtained before vaccine injection.
- PepCan vaccine or placebo (salt water) will be injected under your skin in either one of your arms or one of your legs.
- After resting for at least 30 min after the injection, vital signs will be obtained.
- You'll be offered a dose of ibuprofen or naproxen. You do not have to take it, but it might help limit possible reactions that may occur.
- You will be given a stool collection kit with another questionnaire asking about antibiotic usage, instructions and shipping supplies to send the sample back to UAMS.

## Visit 8 (6 months after Visit 7; UAMS Winthrop P. Rockefeller Cancer Institute)

- You'll be asked if you experienced any side effects or reactions to the last vaccination.
- You'll be asked about any medication changes.


Sponsor: UAMS

- Women of childbearing potential will be asked to take a urine pregnancy test.
- Vital signs will be obtained and a physical exam will be performed.
- You will be asked to swish approximately one tablespoon of mouthwash for at least 30 seconds in your mouth and spit it into a specimen cup. You should not have brushed for 2 hours and eaten for 10 minutes before doing so.
- You will be asked to complete a questionnaire about antibiotic usage.
- Eight to ten tubes of blood (up to 7 tablespoons total) will be drawn for clinical and immunology testing. Additional tubes may be drawn for standard of care.
  - The blood may be used to study how your white cells are reacting to HPV, to allow them to grow in a laboratory, for tissue (HLA) typing, genetic testing of your immune cells and related genes, and other similar tests. In addition, the blood may be used for other testing to see if the vaccine worked in your body by examining proteins and other types of specialized cells.
- You will be given a stool collection kit with another questionnaire asking about antibiotic usage, instructions and shipping supplies to send the sample back to UAMS.

## Visit 9 (6 months after Visit 8; UAMS Winthrop P. Rockefeller Cancer Institute)

- You'll be asked if you experienced any side effects or reactions since the last visit.
- You'll be asked about any medication changes.
- You'll be asked to complete the Visit 9 Questionnaire. It will ask you about your overall experience in the study, whether you would participate in a similar study again, whether you would recommend that others participate in a similar study and whether we may anonymously use any comments you make on the form in publications and other study materials.
- Women of childbearing potential will be asked to take a urine pregnancy test.
- Vital signs will be obtained and a physical exam will be performed.
- Eight to ten tubes of blood (up to 7 tablespoons total) will be drawn for clinical and immunology testing. Additional tubes may be drawn for standard of care.
  - The blood may be used to study how your white cells are reacting to HPV, to allow them to grow in a laboratory, for tissue (HLA) typing, genetic testing of your immune cells and related genes, and other similar tests. In addition, the blood may be used for other testing to see if the vaccine worked in your body by examining proteins and other types of specialized cells.

#### **Optional Follow-Up Visit**

A follow-up visit may be scheduled after the screening visit, after a vaccination visit and at any time during study participation to receive follow-up instructions or to be evaluated for side effects.

#### Recurrence

If you experience recurrence, you will not receive any further study treatment or have any more study visits. You will be asked to fill out the "Recurrence Questionnaire" which will ask you to describe your experience as a participant in the study. You will then have completed the study.


#### Other

- If you experience any significant side effects related to the vaccine (also called "dose-limiting toxicities"), you will be treated for these side effects. You will not receive the remaining vaccine doses; however, your participation in the study will continue. Your visits will remain the same as listed above including the collection of blood, spit, and stool for research.
- The investigator or sponsor may terminate the study at any time without your consent.
- You will be informed of any new significant findings that may affect your willingness to continue in the study.
- Clinically relevant research results, including individual research results, collected during
  the study using standard tests/procedures may be provided to your at your request in
  accordance with UAMS Department of Health Information Management policies and
  requirements. However, research information and results obtained using research-only
  tests are not considered standard-of-care and, therefore, will not be released to you.
- You will not be notified about the results of the study. We may, however, publish the results in an academic journal. (What we publish will not include anything that can identify you.)
- If you withdraw from the study or are withdrawn by the investigator, you will be asked to
  complete an Early Termination Questionnaire. This questionnaire will ask why you are
  leaving the study early, what was your overall experience like, and whether you would
  choose to participate in a similar study in the future or recommend that others participate in
  a similar study.
- You will be notified whether you received PepCan or placebo via e-mail and/or standard mail after the study has completed. This may take several years.

#### **RISKS AND DISCOMFORTS**

#### **Vaccine Injection**

- The possible risks of injection of the study drugs are bleeding, infection, large immune response, pain, and scarring. These risks will be minimized by the presence of licensed medical personnel who will be present during and give the injections. Large local immune reactions of red and puffy skin will be treated with ice pack and a cream that is applied to that area of skin. If a large immune reaction occurs, you will be treated immediately by trained personnel. Any vaccine may potentially cause a life-threatening systemic reaction, rarely resulting in death. The reaction is called anaphylaxis. Anaphylaxis is a sudden, severe, potentially fatal allergic reaction that can involve various areas of the body (such as the skin, respiratory tract, gastrointestinal tract, and cardiovascular system). Symptoms can occur within minutes or up two hours after contact with an allergy-causing substance, but in rare instances may occur up to four hours later. Symptoms of an anaphylactic reaction may begin with a tingling sensation, itching, or metallic taste in the mouth. Other symptoms can include hives, a sensation of warmth, asthma symptoms (shortness of breath and/or wheezing), and swelling of the mouth and throat area.
- Adverse events are undesirable side effects that may occur. Adverse events or risks that
  also may occur include nausea, flu-like syndrome, fever, headache, chills, and muscle
  aches. Most of these side effects can be limited by taking ibuprofen or naproxen with your
  vaccinations. In our earlier preliminary study, the most common reaction seen in most
  vaccine recipients was injection-site reaction (redness, itching, swelling) both immediate
  and delayed (occurring more than 24 hours after injection).
- The possible risks of taking ibuprofen or naproxen are in rare instances: difficulty breathing; swelling of your face, lips, tongue, or throat; and in some people: gastrointestinal problems; rash or other skin problems; kidney problems; or heart problems.

Sponsor: UAMS

- This particular treatment or procedure may involve risks that are unknown at this time.
- This particular treatment or procedure may involve risks, which are currently unforeseeable, to the participant, embryo, or fetus if the participant is or may become pregnant.

#### **Blood Draw**

The risks of drawing blood include temporary discomfort from the needle in your arm, bruising, swelling at the needle site and, in rare instances, infection.

#### **LEGAL RIGHTS**

You do not give up any legal rights to which you are otherwise entitled to by signing the consent form. You may also refuse to participate without loss of benefits.

#### **TREATMENT**

In the event of complications, injury, or illness resulting from your participation in this study, appropriate medical care will be provided. This treatment may include first aid, emergency treatment, and/or follow-up care. This treatment may be billed to you or your insurance company in the normal manner. You will be responsible for any co-pay or deductibles. The principal investigator and this institution have made no provision to reimburse you for the cost of medical care or to pay for any lost wages, pain and suffering, hospitalization, or other expenses you may incur as the result of any such complication, injury or illness. If you develop a medical problem related to the study or have any questions concerning the study, please call Dr. Atig at (501) 686-8530 or after hours at (501) 686-6080.

#### **BENEFITS**

There may be no benefit to you from participating in this research. The intended benefit is the development of a therapeutic vaccine regimen to reduce cancer recurrence for patients with previously diagnosed head and neck cancer. However, the main aim of the study is to examine its safety. Information to be obtained in this study may be of benefit to humankind in the future if it helps to develop a new therapeutic vaccine. The biospecimens and other information from this study may be used for commercial gain; you will not have a share of that income.

#### ALTERNATIVE TREATMENT

If you do not participate in this study, you will still be able to receive the current standard-of-care treatment. Please feel free to talk to your doctor about your choices.

#### REIMBURSEMENT

Travel stipends will be available for Visits 1-9 (except the Screening Visit) as described below. Stipends will be calculated and verified (by study staff) based on mileage from point of origin to the appointment location using internet mapping software, such as Google maps or MapQuest. Stipends will be provided in the form of pre-loaded gift cards.

#### Stipends amounts:

- \$20 per visit for those travelling less than 50 miles
- \$60 per visit for those travelling more than or equal to 50 miles but less than 100 miles
- \$80 per visit for those travelling more than or equal to 100 miles but less than 150 miles
- \$100 per visit for those travelling more than or equal to 150 miles but less than 200 miles
- \$120 per visit for those travelling more than or equal to 200 miles

The maximum amount of gift cards that can be paid per calendar year is limited to \$600. If the amount earned exceeds this limit, the balance will be paid in the next calendar year.

In accordance with the United States IRS tax guidelines, payments paid to an individual per calendar year (January-December), equal to or greater than \$600.00 that are not reimbursements with receipts, are considered income and are taxable. UAMS requires a W-9 to be on file for all clinical trial participants regardless of the amount of payment. If your payments were equal to or greater than \$600.00 in that calendar year, UAMS will send you a 1099-MISC form to file with your taxes. Your name, address, and social security number are needed to process these payments. The 1099-MISC will be sent in January of the following year as required by the IRS. If your payments were not greater than \$600 in the calendar year, you will not receive a 1099-MISC form and you will not have to file this on your taxes.

If you are a recipient of Social Security Income (SSI), Social Security Disability Income (SSDI) recipient, or other income based assistance programs, the additional income from this study will increase your yearly income and possibly making you ineligible for these benefits. If you are currently receiving SSI, Medicaid or Medicare low-income subsidies, please ask your study coordinator for details. Please contact your Social Security Office or your financial advisor if you have any questions.

#### CONFIDENTIALITY

You have a right to privacy. All records are confidential; however, there are risks of loss of confidentiality due to the nature of research. Every effort will be made to keep your information confidential; however, this cannot be guaranteed.

The risks of loss of confidentiality include your information being released to people who are not authorized to access your information. To minimize such an event, your results will be protected and handled as confidentially as possible within the law, including the results of genetic testing, which would reveal a portion of your genetic make-up. All results will be stored and published using codes instead of information that can identify you.

If you are a UAMS patient, you have a UAMS medical record. If you have never been a UAMS patient, a UAMS medical record will be created for the purposes of this study. Results of some research tests and procedures will be included in your UAMS medical record. All information within your medical record can be viewed by individuals authorized to access the record.

Those persons who receive your health information may not be required by Federal privacy laws (such as the Privacy Rule) to protect it and may share your information with others without your permission, if permitted by laws governing them. You do not have to sign this consent form. If you choose not to sign, it will not affect your treatment, payment or enrollment in any health plan or affect your eligibility for benefits. However, you will not be allowed to be a participant in this research study.

By signing this form you are allowing your records (including information that identifies you) to be made available to qualified personnel on Dr. Atiq's study team, and for the FDA, the Office for Human Research Protections, the UAMS IRB, and other institutional oversight offices. The results of this study may be published in a scientific journal or book. Your name or any information to identify you would not be used. Records will be kept regarding your participation in the study. The records will be made available for review only as required by the FDA under the guidelines established by the Federal Privacy Act and the UAMS IRB.

Sponsor: UAMS

Your individual genetic data and health information may be submitted to controlled-access databases. This means that only researchers who apply for and get permission to use the information for a specific research project will be able to access the information. For example, the National Institutes of Health (NIH) has implemented a new database (called the database of Genotypes and Phenotypes) that allows us to submit de-identified genotype (your genetic code) and phenotype (protein produced by your genetic code) data obtained from research associated with your specimen. Although UAMS researchers will not link this research information to your name or other information that could be used to identify you, there is a slight possibility that others could link your DNA in the NIH database with your identity. For example, it would be possible for a person who had your identity and your DNA profile to find your DNA in a Federal Database under the Freedom of Information Act. This would be very rare but could be done by law enforcement, for example. Researchers approved to access information in these databases will agree not to attempt to identify you.

In addition, your information may be submitted to public, unrestricted databases that anyone can use. For example, some public databases include information on large numbers of genetic variations in DNA code; ethnic group and sex; and whether or not individuals have a particular disease. This public information will not be labeled with your name or other information that could be used to identify you easily. However, it is possible that the information from your genome, when combined with information from other public sources could be used to identify you, though we believe it is unlikely that this will happen.

By law, the study team must release certain information to the appropriate authorities if at any time during the study there is concern that abuse has possibly occurred or you disclose a desire to harm yourself or others.

While this study does not specifically test for any communicable diseases, Arkansas law requires certain communicable diseases to be disclosed to the Arkansas Department of Health if they are discovered.

#### HIPAA RESEARCH AUTHORIZATION

As part of the research study in which you are consenting to participate, we need to collect health information that identifies you. We may collect demographic data (such as date of birth, address, social security number for reimbursement purposes), health and medical history (including doctor's notes and clinic records), records from your study visits, and laboratory and test results. We will only collect information that is needed for this research. For you to be included in this research, we need your permission to collect, create, and share this information with the research team.

By signing this form, you are giving us permission to create, collect, use, and share your health information as described above. Your information could be shared with the groups listed above and institutional review committees whose job is to ensure we are protecting your information correctly. Any records or information released might be redisclosed by the person receiving them and will not be covered under the federal privacy laws. Your health information will be kept at least for the durations required by the institutional and federal requirements. Records relating to research conducted under a US FDA IND (21 CFR 312.62(c)) such as this study must be retained for two years after the date a marketing application is approved for the drug for the indication for which it is being investigated; or, if no application is to be filed or if the application is not approved for such indication, for two years after the investigation is discontinued and FDA is notified.

You do not have to sign this form. However, if you decide not to sign this form, you cannot participate in the research study. If you sign this form, but decide later that you no longer want us to collect or share your information, simply send a letter to Dr. Atiq at 4301 West Markham Street, Slot 508, Little Rock, AR 72205. If you do revoke your permission, you cannot continue to participate in the research. However, in order to maintain the reliability of the research, we may still use and share your information that was collected before the principal investigator received your letter withdrawing the permissions granted under this authorization. All clinical information will be available to you as standard of care medical information. Research information collected during the study is not considered standard of care and, therefore, will not be released to you.

This authorization to collect, use, and share your health information does not expire. In addition, you may choose to allow the use of your cell samples for future research. If you make this choice, your authorization will last for the life of the samples, as these will be stored indefinitely until needed for a future research study. If you decide not to sign this form or change your mind later, this will not affect your current or future medical care at UAMS.

#### CONFLICT OF INTEREST DISCLOSURE

This research study is designed to test a product invented by Dr. Nakagawa. UAMS and Dr. Nakagawa are entitled to a share of royalties received from any future sales of this product if it is ultimately approved by the FDA. The financial value of this interest might be affected by the results of this study. This means that UAMS and Dr. Nakagawa could gain or lose money depending on the results of this study.

#### **CLINICALTRIALS.GOV REGISTRY**

This study will be registered with Clinicaltrials.gov. A description of this clinical trial will be available on <a href="http://www.clinicaltrials.gov">http://www.clinicaltrials.gov</a> as required by US Law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this web site at any time.

#### WHETHER OR NOT TO PARTICIPATE

Your participation is VOLUNTARY. You may refuse to participate or decide to withdraw from the study at any time. You may refuse to participate in the study without loss of benefits to which you are otherwise entitled. If you choose to guit the study, there will be no prejudices against you for other studies or care at UAMS. You may stop being part of the study by simply informing Dr. Atiq or a Study Coordinator.

Dr. Atig, or other study investigators (physicians), may terminate your participation in this study at any time after he/she has explained the reasons for doing so. Reasons for termination may include your safety, not following appointment scheduling, or not being able to contact you, among other reasons.

Sponsor: UAMS

#### **GENETIC STUDIES**

As part of this study, white cells from your blood samples may be tested for tissue (HLA) types and immune cell genes, as well as other studies. Your oral and stool samples will be tested to study bacteria and viruses, but your genetic information may also be revealed. The samples will be assigned a number instead of your name. The number will be linked to your name but the code will be stored under lock and key in the laboratory of the principal investigator. You can withdraw your cell sample at any time. If at any time you would like to withdraw your stored sample, please write Dr. Atig at 4301 West Markham Street, Slot 508, Little Rock, AR 72205.

With genetic testing of your tissue, there is a potential risk of loss of confidentiality. Every effort will be made to protect your confidential information, but this cannot be guaranteed. The genetic information obtained as a result of your participation in this research will not be included in your medical record. Information from which you may be personally identified will be maintained in a confidential, secure location in Dr. Nakagawa's (the Sub-Investigator) laboratory, accessible only by authorized members of the study team, and will not be disclosed to third parties except as described in this consent form, with your permission, or as may be required by law.

Genetic testing involves unique risks such as psychological and social risks and the risk of reidentification. Social risks include being stigmatized, discriminated against, labeled, or having difficulty obtaining employment or insurance. Some of your genetic information may be sent to other scientific or commercial databases, such as one maintained by the National Institutes of Health, for other researchers to use. This information would include a code number instead of your name. There is a risk that someone could trace the information back to you. Even without your name or other identifiers, your genetic information is unique to you. We believe the chance that someone will identify you is very small, because your samples will be coded (without your name or identifying information), but the risk may change in the future as people come up with new ways of tracing information. The genetic testing will be done for research purposes only, and we do not plan to return any results to you or your doctor.

The Genetic Information Nondiscrimination Act (GINA) is a Federal law that will protect you in the following ways:

- Health insurance companies and group plans may not request genetic information from this research;
- Health insurance companies and group plans may not use your genetic information when making decisions regarding your eligibility or premiums;
- Employers with 15 or more employees may not use your genetic information when making a decision to hire, promote, or fire you or when setting the terms of your employment.
- GINA does not protect you against genetic discrimination by companies that sell life insurance, disability insurance, or long-term care insurance. GINA also does not protect you against discrimination based on an already-diagnosed genetic condition or disease.

In order to participate in this research study, you need to allow your samples to be tested for the genetic studies mentioned above. If you do NOT agree to allow your samples to be tested for the genetic studies mentioned above, you will not be allowed to participate in this study.

Date

#### **FUTURE USE OF REMAINING SAMPLES**

Printed Name of Person

**Obtaining Consent** 

After we complete our tests, we would like to save any leftover samples for future research studies on HPV. Your blood, cell, oral and stool samples will be frozen and will be stored with a number assigned to them instead of your name. The cell samples may be stored indefinitely until needed for a future research study. The number will be linked to your name, which means you can withdraw your cell sample at any time. If at any time you would like to withdraw your stored sample, please write Dr. Atiq at 4301 West Markham Street, Slot 508, Little Rock, AR 72205.

You may agree to participate in this research study, but refuse to allow your samples to be stored

for future research. Please **initial and date** the appropriate line. Initials: Date: I AGREE to have my leftover samples stored for future research. Initials: \_\_\_\_\_ Date: \_\_\_\_\_ I DO NOT AGREE to have my leftover samples stored for future research. If you do not agree to the use of your leftover samples for future research, they will be taken out of the freezers and will be discarded at the end of this study. Your health information will be kept at least for the durations required by the institutional and federal requirements as noted in the HIPAA section above. **SIGNATURE** I have read the above statements and have been able to ask questions and express concerns, which have been satisfactorily responded to by the study team. I understand the purpose of the study as well as the potential risks and benefits that are involved. I hereby give my informed and free consent to be a participant in this study. I have been told that I will be given a copy of this consent form. MY SIGNATURE INDICATES THAT I ALLOW MY SAMPLES TO BE TESTED FOR GENETIC STUDIES AND HAVE DECIDED TO TAKE PART IN THIS STUDY. Printed Name of Participant Signature Date

Signature